CLINICAL TRIAL: NCT00777621
Title: Caloric Restriction, Exercise, and Glucoregulation in Humans
Acronym: CREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Edward Weiss, Ph.D., Associate Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K01DK080886 (NIH); K01DK080886 (NIH); 1K01DK080886-01 (NIH)
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Caloric Restriction; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calorie restriction (Active Comparator)
  Interventions: Other: Calorie Restriction
- Exercise (Active Comparator)
  Interventions: Other: Exercise
- Calorie restriction and exercise (Experimental)
  Interventions: Other: Calorie Restriction and Exercise

INTERVENTIONS:
Other: Calorie Restriction — This group will undergo a 20% reduction in energy intake without any change in energy expenditure.
  Arms: Calorie restriction
Other: Exercise — This group will undergo a 20% increase in energy expenditure by exercising without any change in energy intake.
  Arms: Exercise
Other: Calorie Restriction and Exercise — This group will undergo 10% reduction in energy intake and a 10% increase in energy expenditure via exercise.
  Arms: Calorie restriction and exercise

SUMMARY:
Weight loss induced by caloric restriction alone (CR) and by exercise alone (EX) result in similar effects on blood glucose and insulin. The purpose of this study is to assess the hypothesis that weight loss through caloric restriction plus exercise will result in greater improvements on glucose tolerance and insulin action than similar weight losses through CR or EX alone.

DETAILED DESCRIPTION:
Participants are randomized into caloric restriction, exercise, and caloric restriction plus exercise weight loss groups. Measurements of blood glucose and insulin, oral glucose tolerance, and matched glucose infusion will be done at baseline and after weight loss of 6% of body weight. Other tests include maximal oxygen uptake (VO2max), strength tests, blood pressure, blood lipids, serum inflammatory markers, dual X-ray absorptiometry (DEXA) for bone density and body composition, physical activity levels, dietary intakes, and measures of arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* females postmenopausal
* no diabetes, cardiovascular disease, cancer
* no orthopedic problems
* not currently exercising
* BMI between 25 and 29.9
* nonsmokers

Exclusion Criteria:

* current regular exercisers
* premenopausal women
* cardiovascular disease, lung disease, cancer, diabetes

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Glucoregulatory function | 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward P Weiss, PhD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Weiss EP, Jordan RC, Frese EM, Albert SG, Villareal DT. Effects of Weight Loss on Lean Mass, Strength, Bone, and Aerobic Capacity. Med Sci Sports Exerc. 2017 Jan;49(1):206-217. doi: 10.1249/MSS.0000000000001074. PMID 27580151
- [Derived] Weiss EP, Albert SG, Reeds DN, Kress KS, McDaniel JL, Klein S, Villareal DT. Effects of matched weight loss from calorie restriction, exercise, or both on cardiovascular disease risk factors: a randomized intervention trial. Am J Clin Nutr. 2016 Sep;104(3):576-86. doi: 10.3945/ajcn.116.131391. Epub 2016 Jul 27. PMID 27465384
- [Derived] Weiss EP, Albert SG, Reeds DN, Kress KS, Ezekiel UR, McDaniel JL, Patterson BW, Klein S, Villareal DT. Calorie Restriction and Matched Weight Loss From Exercise: Independent and Additive Effects on Glucoregulation and the Incretin System in Overweight Women and Men. Diabetes Care. 2015 Jul;38(7):1253-62. doi: 10.2337/dc14-2913. Epub 2015 Apr 15. PMID 25877812